CLINICAL TRIAL: NCT03639454
Title: Effect on Symptomatic Release of Dry Needling on Patients With Biceps Tendinopathy
Brief Title: Dry Needling Treatment for Biceps Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Li-Wei Chou, Minister of Rehabilitation, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH107-REC2-101
Record Dates: First submitted 2018-08-16; First posted 2018-08-21 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2018-08

CONDITIONS: Bicep Tendinitis
Keywords: dry needling; myofascial trigger point; muscle tone
MeSH Terms: interventions — Dry Needling; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): In this arm, the subjects will receive the intervention of DN on Day1, Day2 and Day4, in total 3 treatments and will be arrange to take efficacy two assessment on Day8 and Day15, separately.
  Interventions: Procedure: dry needling
- Transcutaneous Electric Nerve Stimulation (Active Comparator): In this arm, the subjects will receive the intervention of Transcutaneous Electric Nerve Stimulation on Day1, Day2 and Day4, in total 3 treatments and will be arrange to take efficacy two assessment on Day8 and Day15, separately.
  Interventions: Procedure: Transcutaneous electrical nerve stimulation

INTERVENTIONS:
Procedure: dry needling — Dry needling, also known as myofascial trigger point dry needling, is an well-proved technique in alternative medicine similar to acupuncture. It involves the use of either solid filiform needles or hollow-core hypodermic needles for therapy of muscle pain, including pain related to myofascial pain syndrome. Dry needling is sometimes also known as intramuscular stimulation (IMS).
  Arms: Dry needling
Procedure: Transcutaneous electrical nerve stimulation — Transcutaneous electrical nerve stimulation (TENS or TNS) is the use of electric current produced by a device to stimulate the nerves for therapeutic purposes.
  TENS, by definition, covers the complete range of transcutaneously applied currents used for nerve excitation although the term is often used with a more restrictive intent, namely to describe the kind of pulses produced by portable stimulators used to treat pain. The unit is usually connected to the skin using two or more electrodes. A typical battery operated TENS unit is able to modulate pulse width, frequency and intensity. Generally TENS is applied at high frequency (>50 Hz) with an intensity below motor contraction (sensory intensity) or low frequency (<10 Hz) with an intensity that produces motor contraction.
  Arms: Transcutaneous Electric Nerve Stimulation

SUMMARY:
Biceps tendinopathy is a common cause in shoulder-pain symptoms. The major mechanism is overuse of the biceps muscles. The long-term accumulated and poor repaired trauma causes myofascial trigger points in the related muscles.

We will conduct the randomized, single blind experiment to evaluate the immediate, short-term, and long-term effect of DN.

DETAILED DESCRIPTION:
Biceps tendinopathy is a common cause in shoulder-pain symptoms. The major mechanism is overuse of the biceps muscles. The long-term accumulated and poor repaired trauma causes myofascial trigger points in the related muscles. Common symptoms are pain in the anterior shoulders and radiating pain in the biceps. Pain can be further elicited with lifting, pulling and repetitive overhead activity. Therefore, it can have a major impact on the patient's activity of daily life.

The investigator performed dry needle (DN) treatments with acupuncture needles. Stimulating the effected muscle , the investigator move the needle forward and backward several times. Muscle twitch may occur by our procedure. The pain caused by myofascial trigger points can be decreased effective simultaneously. So far, there is no solid research or clinical trial to evaluate the efficacy of the treatment yet.

The investigator will conduct the randomized, single blind experiment to evaluate the immediate, short-term, and long-term effect of DN. Outcome measures include visual analog scale, shoulder pain and disability index, pressure pain threshold, pain-free grip test, muscle tone changes and ultrasonographic evaluation of biceps peritendinous effusion.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects older than 20 years of age who can cooperate with the experimental volunteers.
2. Suffering from biceps tendon lesions for more than one month, and subjective pain intensity (VAS) greater than 5 points.
3. There is a local tender point in front of the shoulder, and the shoulder joint pronation test can induce pain.
4. Under soft tissue ultrasound, the thickness of Biceps Peritendinous Effusion (BPE) on the affected side of the biceps tendon is greater than 1 mm.

Exclusion Criteria:

1. There are contraindications to general treatment, such as serious medical problems, recent serious trauma, or pregnant women.
2. There has been a history of drug abuse (including excess alcohol) that affects pain assessors.
3. Have received shoulder, neck or upper back surgery.
4. People with central or peripheral nerve disease.
5. Cognitive impairment, unable to cooperate with the experimenter.
6. Patients currently receiving other treatments for Biceps tendinopathy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scales | 1 day
  The visual analogue scale or visual analog scale is a psychometric response scale which can be used in questionnaires. This tool used to help a person rate the intensity of certain sensations and feelings, such as pain. A straight line of 100mm is actually marked with 0 mm on the far left and 100mm on the far right. Two faces are drawn on both ends. Explain to the patient that 0 mm means no pain and 100 mm means very painful. From the left end The right shift indicates more and more pain. Take a pen and let the patient draw a short line vertically on the line, representing his painful position, and record the measured cm value. In this test, if the score of the subject decreases, it can represent the treatment is helpful for the improvement of the patient's pain.

SECONDARY OUTCOMES:
Pressure Pain Threshold | 1 day
  Pressure pain threshold (PPT) is defined as the minimum force applied which induces pain. This measure has proven to be commonly useful in evaluating tenderness symptom.
Muscle tension | 1 day
  Muscle tension is the muscle's resistance to passive stretch during resting state. The measuring tool called Myotone will calculate three parameters such as tone, elasticity and stiffness and get a value to represent the muscle tension. If the value decrease, it can represent the treatment is helpful for the subjective muscle relax.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Chou, PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen IW, Liao YT, Tseng H, Lin HC, Chou LW. Pain, function and peritendinous effusion improvement after dry needling in patients with long head of biceps brachii tendinopathy: a single-blind randomized clinical trial. Ann Med. 2024 Dec;56(1):2391528. doi: 10.1080/07853890.2024.2391528. Epub 2024 Aug 14. PMID 39140690